CLINICAL TRIAL: NCT06445283
Title: Determination of Venous Thromboembolism Risk and Nursing Practices in Patients Hospitalized in Medical Services in a Tertiary University Hospital: Point Prevalence Study
Brief Title: Determination of Venous Thromboembolism Risk and Nursing Practices in Patients Hospitalized in Medical Services
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Humeyra Zengin, RN,PhD, Director of Nursing Services, Hacettepe University
Other Study IDs: HU-NS-VTERisk001
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Venous Thromboembolism
Keywords: Venous Thromboembolism; Nursing Practise
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Determination of VTE risk levels — Determination of VTE risk levels of patients using IMPROVE risk assessment tool according to deep vein thrombosis and pulmonary embolism risk factors

SUMMARY:
Together with individual predisposition to form vascular clots and clinical conditions that further increase this risk, venous thromboembolism (VTE) poses a significant additional morbidity and mortality risk for the majority of the world's population. Although VTE causes serious disability and death when undiagnosed, it is a medical condition that can be prevented when diagnosed early. Although all hospitalized patients are at risk of DVT, studies have shown that 75% of hospitalized patients are hospitalized in internal clinics.As a result of this observational study, it was aimed to determine the VTE risk levels of the patients from the time of hospitalization and to determine preventive nursing care for VTE.

DETAILED DESCRIPTION:
Venous Thromboembolism (VTE) refers to interrelated diagnoses such as Deep Vein Thrombosis (DVT) and Pulmonary Embolism (PE). 10-20% of venous thromboembolic events occur in medical patients and 10-80% in intensive care patients. Recognized as a major complication for medical and surgical patients, VTE has been described as the 'silent killer' of hospitalized patients. During the Covid-19 pandemic in recent years, high rates of thrombolytic events have been reported in hospitalized COVID-19 patients. Nurses have an important role in identifying risk factors for VTE, taking precautions and assessing patient compliance with these precautions. The nurse should identify risk factors in the preoperative period, long-term and intensive care hospitalizations by taking a comprehensive history and physical assessment of the patient before hospitalization. There are several risk assessment models developed to assess the risk of VTE for application to inpatient medical patients. There are various risk assessment models developed for application to inpatient medical patients. Padua and IMPROVE VTE risk assessment models are frequently used. In the literature, it is stated that the Padua model gives moderate results and the IMPROVE model gives moderate-good results in predicting risk (1). Therefore, risk levels were not determined with the IMPROVE risk assessment tool in this study.

ELIGIBILITY:
Inclusion Criteria:

* To be conscious,
* Consent of the patient's relatives to participate in the study in unconscious patients
* 24 hours have passed since hospitalization
* The patient admitted to hospitalization has been pre-assessed by the nurse and the pre-assessment form and nurse observation form have been completed

Exclusion Criteria:

* Surgical patients
* Pregnant patients
* Refusing to participate in the study during the completion of the data collection forms.
* In unconscious patients, the patient's relatives did not give consent to participate in the study
* Unconscious patient whose relatives cannot be reached
* The patient admitted to hospitalization was not pre-assessed by the nurse and the pre-assessment form and nurse observation form were not filled out

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the study will consist of patients hospitalized in the medical clinics of an Adult Hospital of a University. The Adult Hospital serving adult patients has a capacity of 801 beds and the number of beds allocated for medical services is 211.
Sampling Method: Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Determination of IMPROVE risk model risk levels according to deep vein thrombosis and pulmonary embolism risk factors | 21 February 2024
  IMPROVE VTE Risk modeli,the seven risk factors evaluated in this model are history of VTE, thrombophilia, cancer in remission within the last 5 years, lower extremity paralysis or paresthesia (leg falling to the bed within 5 seconds), immobilization (complete immobility in bed or chair for ≥ 1 day), ICU (ICU)/Coronary ICU hospitalization, Age ≥ 60 years. In this model with a maximum of 12 points; 0-1 point range is defined as low VTE risk, 2-3 point range as moderate VTE risk and 4 points and above high VTE risk,

SECONDARY OUTCOMES:
Rate of implementation of nursing practices for VTE risk | 21 February 2024
  Nursing Practise; Informing patients about VTE, To Mobilize the Patient Leg exercises in bed Compression Elastic Socks Intermittent Pneumatic Compression Evaluation of the lower extremities (calf pain, edema, discoloration, tenderness, temperature increase and pulse control, etc.) Daily monitoring of laboratory tests Evaluation of the Glasgow Coma Scale

CONTACTS AND LOCATIONS:
Overall Officials: Humeyra Zengin, Principal Investigator — Director of Nursing Services
Locations (2):
- Turkey (Türkiye) (2):
  - Hacettepe University, Altındağ, Ankara
  - Hacettepe Uviversity, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Skeik N, Westergard E. Recommendations for VTE Prophylaxis in Medically Ill Patients. Ann Vasc Dis. 2020 Mar 25;13(1):38-44. doi: 10.3400/avd.ra.19-00115. PMID 32273920